CLINICAL TRIAL: NCT06194123
Title: Effect of Whitening Agent With Emulsion Gel in Saliva and Halitosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4475
Record Dates: First submitted 2023-12-11; First posted 2024-01-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Xerostomia; Halitosis
MeSH Terms: conditions — Xerostomia; Halitosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): All subjects will be instructed to use the Crest Daily Whitening Serum for 1 week as described on the label. This product is available for purchase at any pharmacy.
  Interventions: Other: Crest Daily Whitening Serum

INTERVENTIONS:
Other: Crest Daily Whitening Serum — one week's use of Crest Daily Whitening Serum as described on the label.

SUMMARY:
The objective of this study is to evaluate how well the study product, Crest Daily Whitening Serum, alleviates Xerostomia and perceived halitosis over 1 week of use.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Can produce an unstimulated salivary flow rate of 0.18mL/min. or less.
* Score of 3 or more on question 1 of the VAS dry mouth scale (How severe is your dryness right now?), evaluated in the Pre-Product Use Dry Mouth & Sensitivity Questionnaire.
* Evidence of currently taking a stable dose (3 months or more) of Xerostomia-inducing medication such as, antihypertensives, anti-anxiety agents, psychiatric remedies, antihistamines and etc.

  • At screening, participants may present the prescription bottle, a picture of the prescriptions bottle or medical records showing the prescription.
* Subject not currently using any teeth whitening or desensitizing products that contain potassium nitrate such as Sensodyne, Pronamel etc.
* Subject willing to comply with the study regimen and products.

  * Not consume alcohol for 24 hours prior to their visit.
  * Not brush their teeth for 1.5 hours prior to their visit.
  * Not have had anything to eat or drink (including chewing gum or eating candy) for 1.5 hours prior to their visit). Water is acceptable to drink up to 1 hour prior to the study visit.
  * Not smoke 1.5 hours prior to their visit

Exclusion Criteria:

i. Subjects who are currently pregnant (self-reported). ii. Unstimulated salivary flow rate of more than 0.18mL/min iii. Subjects that have ever received therapeutic radiation in the head and neck area.

iv. Subjects with a diagnosis of conditions that would affect salivary flow such as Sjogren's Syndrome per the investigator's expert opinion.

v. Subjects with a condition the investigator believes not suitable for the study, such as autoimmune diseases and radiation therapy to head and neck region that impact salivary flow.

vi. Subjects that currently use whitening toothpaste, desensitizing toothpaste, or any other products causing similar results.

vii. Subjects currently participating in any other research studies. viii. Subject unable to provide consent (e.g. Cognitively impaired adults). ix. Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective 1- Visual Analogue Scale for Perceived Dry Mouth | 5, 30, 60 minute post application of product as well as degree of change after a 7 day period of use.
  To observe presence and degree of reduction in the self-reported subjective perception of dryness in the oral cavity at different time intervals after the application of a Whitening Agent with Emulsion Gel in Xerostomic Population

SECONDARY OUTCOMES:
Objective 2- Visual Analogue Scale for Perceived Bad Breath and Saliva Production Increase | 60 minutes post application as well as degree of change after a 7 day period of use.
  To measure presence and degree of reduction of self-reported bad breath and subject's objective measurement of how well saliva production improved on a 1-10 scale at different time intervals with a Whitening Agent with Emulsion Gel in Xerostomic Population

CONTACTS AND LOCATIONS:
Overall Officials: Mabi Singh, DMD,MS, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collins LM, Dawes C. The surface area of the adult human mouth and thickness of the salivary film covering the teeth and oral mucosa. J Dent Res. 1987 Aug;66(8):1300-2. doi: 10.1177/00220345870660080201. PMID 3476596
- [Background] Osailan S, Pramanik R, Shirodaria S, Challacombe SJ, Proctor GB. Investigating the relationship between hyposalivation and mucosal wetness. Oral Dis. 2011 Jan;17(1):109-14. doi: 10.1111/j.1601-0825.2010.01715.x. Epub 2010 Oct 28. PMID 21029258
- [Background] Pramanik R, Osailan SM, Challacombe SJ, Urquhart D, Proctor GB. Protein and mucin retention on oral mucosal surfaces in dry mouth patients. Eur J Oral Sci. 2010 Jun;118(3):245-53. doi: 10.1111/j.1600-0722.2010.00728.x. PMID 20572857
- [Background] Murray Thomson W, Poulton R, Mark Broadbent J, Al-Kubaisy S. Xerostomia and medications among 32-year-olds. Acta Odontol Scand. 2006 Aug;64(4):249-54. doi: 10.1080/00016350600633243. PMID 16829502
- [Background] Thomson WM. Issues in the epidemiological investigation of dry mouth. Gerodontology. 2005 Jun;22(2):65-76. doi: 10.1111/j.1741-2358.2005.00058.x. PMID 15934347
- [Background] Guggenheimer J, Moore PA. Xerostomia: etiology, recognition and treatment. J Am Dent Assoc. 2003 Jan;134(1):61-9; quiz 118-9. doi: 10.14219/jada.archive.2003.0018. PMID 12555958
- [Background] Apperley O, Medlicott N, Rich A, Hanning S, Huckabee ML. A clinical trial of a novel emulsion for potential use as a saliva substitute in patients with radiation-induced xerostomia. J Oral Rehabil. 2017 Nov;44(11):889-895. doi: 10.1111/joor.12545. Epub 2017 Aug 20. PMID 28741683